CLINICAL TRIAL: NCT00043719
Title: Prevention of Postmenopausal Bone Loss With Nitric Oxide
Brief Title: Nitroglycerin Ointment for Preventing Bone Loss in Postmenopausal Women
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sunil J. Wimalawansa , MD, PhD, UMDNJ - Robert Wood Johnson Medical School, Division of Endocrinology
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: R01AR048679 (NIH); NIAMS-069; NOVEL
Record Dates: First submitted 2002-08-12; First posted 2002-08-14 (Estimated); Last update posted 2009-02-02 (Estimated); Status verified 2009-01

CONDITIONS: Osteoporosis; Osteopenia
Keywords: Human Female; Osteoporosis; Postmenopausal; Nitric Oxide; Nitroglycerin; Calcium; Vitamin D
MeSH Terms: conditions — Osteoporosis; Bone Diseases, Metabolic | interventions — Vitamin D

INTERVENTIONS:
Drug: Nitroglycerin ointment
Drug: Calcium supplement with vitamin D

SUMMARY:
Osteopenia and osteoporosis cause thinning of bone tissue and loss of bone density over time. The purpose of this study is to determine the safety and effectiveness of nitroglycerin ointment for the treatment of osteopenia in postmenopausal women.

Study hypothesis: On average, participants in the base therapy cohort who receive placebo ointment control and calcium/vitamin D will lose more bone density than participants in the nitroglycerin cohort over the 36-month period.

DETAILED DESCRIPTION:
Imbalance in the activities of osteoclasts (cells responsible for bone loss) and osteoblasts (cells responsible for bone formation) may lead to fractures, osteopenia, and osteoporosis in postmenopausal women. During postmenopause, decreased estrogen levels and decreased nitric oxide production occur; estrogen replacement therapy has been shown to restore serum nitric oxide levels to normal. Reversing nitric oxide deficiency by using nitroglycerin may prevent further bone loss. The Nitroglycerin as an Option: Value in Early Bone Loss (NOVEL) study will test the safety and efficacy of nitroglycerin ointment for the treatment of osteopenia in postmenopausal women.

Patients will be enrolled in the study for 3 years and will be randomly assigned to one of two groups. The first group will receive nitroglycerin ointment, while the second group will receive placebo ointment. All patients will be given a calcium supplement with vitamin D to be taken daily, and will be instructed to rub the given ointment on their skin daily. Study visits will occur at Month 2 and every six months after Month 2. Phone interviews will be conducted with patients every 2 months throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal for a minimum of 13 months
* Lumbar spine T-score of 0 to -2.5 (0 to -2.0 if over 60 years old) by Dual Energy X-ray Absorptiometry (DEXA) (i.e., evidence of normal bone mass or osteopenia)
* Body Mass Index (BMI) between 18 and 32
* Planning to live in the greater New Brunswick, NJ, area for at least 3 years

Exclusion Criteria:

* Radiographically or DEXA-morphometrically proven vertebral or hip fracture
* Conditions requiring routine use of sublingual, transdermal, or oral nitrates
* Significant postmenopausal symptoms that require estrogen therapy
* Metabolic bone diseases other than postmenopausal bone loss (e.g., active hyperthyroidism, hyperparathyroidism, Paget's disease of bone, etc.)
* Insulin-dependent diabetes mellitus
* Significant migraine headaches
* History of renal calculi
* Cancer within 5 years prior to study entry
* Any condition causing an anticipated life expectancy of less than 3 years
* Failure to maintain 75% to 125% compliance with open-label calcium with vitamin D regimen during the screening period

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200
Dates: Start 2002-07; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
DXA-measured BMD (bone mineral density) of lumbar vertebrae (L2 to L4)

SECONDARY OUTCOMES:
DXA-measured BMD of dual hips (Ward's triangle, femoral neck, and trochanter)
serum osteocalcin
BS-ALP
serum N-telopeptide

CONTACTS AND LOCATIONS:
Overall Officials: Sunil J. Wimalawansa, MD, PhD, Principal Investigator — UMDNJ - Robert Wood Johnson Medical School, Division of Endocrinology
Locations (1):
- UMDNJ-Robert Wood Johnson Medical School, Department of Medicine, Division of Endocrinology, New Brunswick, New Jersey, United States